CLINICAL TRIAL: NCT04771000
Title: A Randomised, Double-blind, Placebo-controlled Trial to Evaluate the Efficacy and Safety of Ambrisentan in Patients With Severe COVID-19
Brief Title: A Study of Micro Dose Ambrisentan in Hospitalized Patients With Respiratory Insufficiency Due to COVID-19
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of recruitment
Sponsor: Noorik Biopharmaceuticals AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: N-003-CRD008
Record Dates: First submitted 2021-02-24; First posted 2021-02-25 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Covid19; Hypoxemia
Keywords: Covid19; Hypoxemia; Endothelin; Endothelin receptor antagonist; Ambrisentan; Micro-dose; Acute Respiratory Distress Syndrome (ARDS); Mechanical ventilation; Pulmonary vasodilator; Hypoxic respiratory failure; Respiratory Failure
MeSH Terms: conditions — COVID-19; Hypoxia; Respiratory Distress Syndrome; Respiratory Insufficiency | interventions — ambrisentan; Propylene Glycol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ambrisentan (Experimental): Ambrisentan, 125µg twice a day for up to 28 days
  Interventions: Drug: Ambrisentan
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ambrisentan — Endothelin receptor antagonist
  Other Names: N-003 (ambrisentan solution)
  Arms: Ambrisentan
Drug: Placebo — Placebo
  Other Names: Propylene glycol
  Arms: Placebo

SUMMARY:
Patients with COVID-19 frequently develop lower respiratory complications. Difficulty breathing and a low concentration of oxygen in the blood are of concern in patients with COVID-19, as they indicate that the lungs may be significantly affected. In some patients, respiratory symptoms may progress to the point where oxygen support is needed (i.e. use of an oxygen prongs, mask or ventilator).

The exact mechanism of why patients with COVID-19 develop low concentrations of oxygen in blood is not fully understood. Some data suggest that the Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2), the virus causing Coronavirus Disease 2019 (COVID-19), can affect the body's blood vessels directly and extensively. In the lung, blood vessels participate in the absorption of oxygen.

Endothelin is a potent hormone produced by human blood vessels. When increased, endothelin can result in the narrowing of blood vessels in the lung and decrease the volume of blood flowing through the lungs. This decrease in in blood flow through the lungs may be one of many factors affecting normal lung function. Ambrisentan can block the effects of endothelin in the body, and this could theoretically improve blood flow through the lungs.

This study will evaluate whether ambrisentan, by blocking the effects of the hormone endothelin in the lungs, improves the breathing capacity of patients with COVID-19, increases the concentration of oxygen in the blood and prevents the progression to respiratory failure and death. Ambrisentan is a drug that is currently used to treat patients with pulmonary hypertension, a disease where blood flow through the lungs is decreased.

Subjects participating in this study are those patients hospitalised with severe respiratory symptoms related to COVID-19, and are considered to be at high-risk of developing respiratory complications. Ambrisentan will be administered in the hospital, and will be continued at home for up to 28 days. In this study, ambrisentan will be administered at much lower doses that those used in patients with pulmonary hypertension.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, multi-centre trial to evaluate the safety and efficacy of ambrisentan for the treatment of severe COVID-19. The population consists of hospitalized subjects who have a confirmed SARS-CoV-2 (a coronavirus (CoV) ) infection, are at high-risk of progression to respiratory failure or death and have low oxygen saturation and/or require oxygen supplementation at the time of admission. Pregnant or lactating women will not be allowed to participate in this study given the teratogenic potential of ambrisentan. Subjects requiring mechanical ventilation or intubation at the time of enrolment are considered to have respiratory failure and will not be allowed into the study, as one primary objective of the study is to evaluate the effect of ambrisentan in preventing respiratory failure.

Enrolled subjects will be randomly assigned to the treatment arm or control arm at a 1:1 ratio. In the treatment arm, subjects will receive ambrisentan on top of the standard-of-care. In the control arm, subjects will receive the administration vehicle only (i.e., placebo) and on top of the standard of care. The study medication (ambrisentan or placebo) will be administered for up to 28 days. In the event that the subject is discharged between Day 4 and Day 28, the subject will continue the study treatment at home until completion of the 28-day study medication regimen. Investigators, the Sponsor and the subject will be blinded to the treatment assignment. A Drug Safety Monitoring Board will be monitoring the safety of the study.

ELIGIBILITY:
Inclusion Criteria:

* Subject (or legally authorized representative) provides informed consent (written or oral) prior to initiation of any study procedures.
* Male or non-pregnant, non-lactating female. Women of child-bearing potential must have a confirmed negative serum pregnancy test at the time of screening and must use a highly effective contraceptive method throughout the study (such as implants, injectables, hormonal contraceptives and condom, double barrier contraception [i.e., condom + diaphragm/spermicidal gel or foam]) and until one month after completing treatment with the study medication. In the case of hormonal contraception, women should have been on a stable regimen for a minimum of three months before study enrolment. Women not of child-bearing potential include post-menopausal females (defined as having a history of amenorrhea for at least one year) or a documented status as being surgically sterile (hysterectomy, bilateral oophorectomy, tubal ligation/salpingectomy). Men must use an effective contraception method (i.e., condom + diaphragm/spermicidal gel or foam, or vasectomy), and should not donate semen during the study. Men are considered to be fertile from the time of puberty, except for those men with permanent sterility secondary to bilateral orchiectomy.
* At least 18 years of age and not older than 85 years of age at time of enrolment
* Confirmed SARS-CoV-2 infection defined as: Positive Real-Time Polymerase Chain Reaction (RT-PCR) result in sample collected in the 10 days prior to randomisation, OR positive antigenic test result in sample collected in the 10 days prior to randomisation.
* Radiological confirmation of pneumonia.
* Subject receiving low-flow oxzgen supplementation of at least 2 L/min and not more than 15 L/min.
* Subject (or legally authorized representative) understands and agrees to comply with planned study procedures.
* Subject (or legally authorized representative) agrees to not participate in any other clinical trial, including clinical trials for the treatment or prevention of COVID-19 or SARS-CoV-2 through Day 30.

Exclusion Criteria:

* Subject at a high risk of death, according to investigator's opinion, in the 3 months following enrollment from other causes than Acute Respiratory Distress Syndrome (e.g., severe neurological damage or cancer patients in terminal stages of the disease).
* Subject currently being treated with an endothelin receptor antagonist.
* Subject currently being treated with another pulmonary vasodilator.
* Anticipated need for high-flow oxygen supplementation, non-invasive mechanical ventilation, endotracheal intubation or tracheostomy at the time of screening.
* History of mechanical ventilation (invasive or non-invasive) in the last 7 days.
* Documented history of end-stage liver disease, cirrhosis or idiopathic pulmonary fibrosis (IPF) with or without pulmonary arterial hypertension.
* Aspartate Aminotransferase (AST) or Alanine Aminotransferase (ALT) > 3-times the upper limit of normal (ULN).
* Anticipated discharge from the hospital or transfer to another hospital which is not a study site within 96 hours.
* Participation in another interventional clinical trial in the 15 days prior to enrollment.
* Known hypersensitivity to ambrisentan or propylene glycol.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2021-02-08 (Actual); Primary Completion 2023-02-27 (Actual); Study Completion 2023-02-27 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects alive and not having developed respiratory failure from randomization to Day 14 | 30 days
  The number of patients that are alive and have not developed respiratory failure by day 30 after entering the study will be compared between the experimental and placebo arms

SECONDARY OUTCOMES:
Proportion of subjects alive and free of respiratory failure at Day 14 and Day 30 | 14 days and 30 days
  The number of patients that are alive and have not developed respiratory failure on day 14 will will be compared between the experimental and placebo arms
Proportion of subjects alive and not requiring oxygen supplementation or higher respiratory support at Day 14. | 14 days
  The number of patients not requiring supplemental oxygen, or any other type of respiratory support at day 14 will be compared between the experimental and placebo arms
Time to hospital discharge (up to Day 30) | 30 days
  The time in days required for subjects to be discharged from the first hospitalisation will be estimated and compared between the experimental and placebo groups
Proportion of subjects admitted to the Intensive Care Unit or High-Dependency Unit (up to Day 30) | 30 days
  The number of patients who qualified for admission or where admitted to an intensive care or a high-dependency unit at any time during the first 30 days after entering the study will be estimated and compared between the experimental and placebo groups
Time until weaning from oxygen therapy (up to Day 30) | 30 days
  The time in days subjects required to breathe independently and without oxygen support will be estimated and compared for the experimental and placebo groups
Time until weaning from respiratory support other than low-flow oxygen supplementation for subjects having developed respiratory failure (up to Day 30) | 30 days
  The time in days subjects required to breathe independently with or without supplemental oxygen will be estimated and compared for the experimental and placebo groups
Change in SpO2/FiO2 from baseline to the time-weighted average obtained on Day 3 | 3 days
  The difference in blood oxygen saturation (SpO2) corrected by the inspired fraction of oxygen (FiO2) between baseline and the time-adjusted average calculated for day 3 will be compared between the experimental and placebo arms
Change in SpO2/FiO2 from baseline to the time-weighted average obtained on Day 1 | 1 day
  The difference in blood oxygen saturation corrected by the inspired fraction of oxygen between baseline and the time-adjusted average calculated for day 1 will be compared between the experimental and placebo arms
Change in SpO2/FiO2 from baseline to the time-weighted average obtained on Day 2 | 2 days
  The difference in blood oxygen saturation corrected by the inspired fraction of oxygen between baseline and the time-adjusted average calculated for day 2 will be compared between the experimental and placebo arms
Proportion of subjects experiencing at least one event of venous thrombosis (specifically deep venous thrombosis or pulmonary embolism) (up to Day 30). | 30 days
  The number of patients who developed thrombosis or pulmonary embolism during the first 30 days after entering the study will be estimated and compared between the experimental and placebo groups
Proportion of subjects by clinical status reported on a 11-point ordinal scale at Day 14 and Day 30 | 14 days and 30 days
  The number of patients classified according to an 11-pont scale on their clinical status at day 14 and day 30 will be calculated and compared between the experimental and placebo groups. The 11-point scale is as follows: Uninfected (0 points), Ambulatory and Asymptomatic (1 point), Symptomatic and independent (2 points), Symptomatic requiring assistance (3 points), Hospitalized with no oxygen therapy (4 points), Hospitalized with oxygen by mask or nasal prongs (5 points), Hospitalized with oxygen by non-invasive ventilation or high flow (6 points), Intubation and mechanical ventilation, PaO2/FiO2 ≥ 150 or SpO2/FiO2 ≥ 200 (7 points), Mechanical ventilation, PaO2/FiO2 <150 (SpO2/FiO2 < 200) or vasopressors (8 points), Mechanical ventilation, PaO2/FiO2 < 150 (SpO2/FiO2 < 200) and vasopressors, dialysis or Extracorporeal Membrane Oxygenation (ECMO) (9 points), Dead (10 points).
Time to death due to any cause (up to Day 30) | 30 days
  For those subjects dying in the first 30 days after study entry, the time from study entry to death will be estimated and compared between the experimental and placebo groups
All-cause mortality at Day 30 | 30 days
  The number of patients dying during the study observation period independent of the cause of death will be calculated and compared between the experimental and placebo groups.

OTHER OUTCOMES:
Change in SpO2/FiO2 from baseline to the time-weighted average obtained on Day 14 | 14 days
  The difference in blood oxygen saturation corrected by the inspired fraction of oxygen between baseline and the time-adjusted average calculated for day 14 will be compared between the experimental and placebo arms

CONTACTS AND LOCATIONS:
Overall Officials: Rok Civljak, MD, Principal Investigator — University Hospital for Infectious Diseases Fran Mihaljevic
Locations (13):
- Croatia (2):
  - General Hopital Zadar, Zadar
  - University Hospital for Infectious Diseases Fran Mihaljevic, Zagreb
- Spain (11):
  - Hospital Universitario Virgen de las Nieves, Granada, Comunidad de Andalucia
  - Hospital Universitario San Cecilio, Granada, Comunidad de Andalucia
  - Hospital Universitario de Jaén, Jaén, Comunidad de Andalucía
  - Hospital Universitario de Galdakao-Usansolo, Galdakao, Comunidad de Bizkaia
  - Complejo Hospitalario de Navarra, Pamplona, Comunidad de Navarra
  - Hospital Rey Juan Carlos, Móstoles, Madrid
  - Hospital Universitario de Cabueñes, Gijón, Principality of Asturias
  - Hospital Universitario Infanta Leonor, Madrid
  - University Hospital 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital de Emergencias Enfermera Isabel Zendal, Madrid

IPD SHARING:
Plan to Share IPD: Undecided
Not yet discussed or decided

REFERENCES:
- [Background] Argulian E, Sud K, Vogel B, Bohra C, Garg VP, Talebi S, Lerakis S, Narula J. Right Ventricular Dilation in Hospitalized Patients With COVID-19 Infection. JACC Cardiovasc Imaging. 2020 Nov;13(11):2459-2461. doi: 10.1016/j.jcmg.2020.05.010. Epub 2020 May 15. No abstract available. PMID 32426088
- [Background] Fox SE, Akmatbekov A, Harbert JL, Li G, Quincy Brown J, Vander Heide RS. Pulmonary and cardiac pathology in African American patients with COVID-19: an autopsy series from New Orleans. Lancet Respir Med. 2020 Jul;8(7):681-686. doi: 10.1016/S2213-2600(20)30243-5. Epub 2020 May 27. PMID 32473124
- [Background] Santamarina MG, Boisier D, Contreras R, Baque M, Volpacchio M, Beddings I. COVID-19: a hypothesis regarding the ventilation-perfusion mismatch. Crit Care. 2020 Jul 6;24(1):395. doi: 10.1186/s13054-020-03125-9. No abstract available. PMID 32631389
- [Background] Gattinoni L, Chiumello D, Caironi P, Busana M, Romitti F, Brazzi L, Camporota L. COVID-19 pneumonia: different respiratory treatments for different phenotypes? Intensive Care Med. 2020 Jun;46(6):1099-1102. doi: 10.1007/s00134-020-06033-2. Epub 2020 Apr 14. No abstract available. PMID 32291463
- [Background] Zhou F, Yu T, Du R, Fan G, Liu Y, Liu Z, Xiang J, Wang Y, Song B, Gu X, Guan L, Wei Y, Li H, Wu X, Xu J, Tu S, Zhang Y, Chen H, Cao B. Clinical course and risk factors for mortality of adult inpatients with COVID-19 in Wuhan, China: a retrospective cohort study. Lancet. 2020 Mar 28;395(10229):1054-1062. doi: 10.1016/S0140-6736(20)30566-3. Epub 2020 Mar 11. PMID 32171076
- [Background] Ackermann M, Verleden SE, Kuehnel M, Haverich A, Welte T, Laenger F, Vanstapel A, Werlein C, Stark H, Tzankov A, Li WW, Li VW, Mentzer SJ, Jonigk D. Pulmonary Vascular Endothelialitis, Thrombosis, and Angiogenesis in Covid-19. N Engl J Med. 2020 Jul 9;383(2):120-128. doi: 10.1056/NEJMoa2015432. Epub 2020 May 21. PMID 32437596
- [Background] Varga Z, Flammer AJ, Steiger P, Haberecker M, Andermatt R, Zinkernagel AS, Mehra MR, Schuepbach RA, Ruschitzka F, Moch H. Endothelial cell infection and endotheliitis in COVID-19. Lancet. 2020 May 2;395(10234):1417-1418. doi: 10.1016/S0140-6736(20)30937-5. Epub 2020 Apr 21. No abstract available. PMID 32325026
- [Background] Kalk P, Senf P, Deja M, Petersen B, Busch T, Bauer C, Boemke W, Kaisers U, Hocher B. Inhalation of an endothelin receptor A antagonist attenuates pulmonary inflammation in experimental acute lung injury. Can J Physiol Pharmacol. 2008 Aug;86(8):511-5. doi: 10.1139/Y08-046. PMID 18758498
- [Background] Deja M, Busch T, Wolf S, Donaubauer B, Petersen B, Skomrock J, Boemke W, Kaisers U. Inhalation of the endothelin-A receptor antagonist LU-135252 at various doses in experimental acute lung injury. J Cardiovasc Pharmacol. 2004 Nov;44 Suppl 1:S151-5. doi: 10.1097/01.fjc.0000166261.42723.b7. PMID 15838267
- [Background] Comellas AP, Briva A. Role of endothelin-1 in acute lung injury. Transl Res. 2009 Jun;153(6):263-71. doi: 10.1016/j.trsl.2009.02.007. Epub 2009 Mar 20. PMID 19446279
- [Background] Henry PJ. Respiratory viral infections and the endothelin system. Pulm Pharmacol Ther. 1998 Apr-Jun;11(2-3):133-40. doi: 10.1006/pupt.1998.0127. No abstract available. PMID 9918745
- [Background] Carpenter TC, Reeves JT, Durmowicz AG. Viral respiratory infection increases susceptibility of young rats to hypoxia-induced pulmonary edema. J Appl Physiol (1985). 1998 Mar;84(3):1048-54. doi: 10.1152/jappl.1998.84.3.1048. PMID 9480968
- [Background] Carpenter TC, Stenmark KR. Endothelin receptor blockade decreases lung water in young rats exposed to viral infection and hypoxia. Am J Physiol Lung Cell Mol Physiol. 2000 Sep;279(3):L547-54. doi: 10.1152/ajplung.2000.279.3.L547. PMID 10956630
- [Background] Oparil S, Chen SJ, Meng QC, Elton TS, Yano M, Chen YF. Endothelin-A receptor antagonist prevents acute hypoxia-induced pulmonary hypertension in the rat. Am J Physiol. 1995 Jan;268(1 Pt 1):L95-100. doi: 10.1152/ajplung.1995.268.1.L95. PMID 7840234
- [Background] Maguire JJ, Kuc RE, Davenport AP. Defining the affinity and receptor sub-type selectivity of four classes of endothelin antagonists in clinically relevant human cardiovascular tissues. Life Sci. 2012 Oct 15;91(13-14):681-6. doi: 10.1016/j.lfs.2012.05.008. Epub 2012 May 23. PMID 22634326
- [Background] Yanagisawa M, Kurihara H, Kimura S, Goto K, Masaki T. A novel peptide vasoconstrictor, endothelin, is produced by vascular endothelium and modulates smooth muscle Ca2+ channels. J Hypertens Suppl. 1988 Dec;6(4):S188-91. doi: 10.1097/00004872-198812040-00056. PMID 2853725